CLINICAL TRIAL: NCT04408560
Title: Evaluation of the Efficacy of a Homeopathic Protocol to Reduce the Onset or Aggravation of Joint Pain or Stiffness Following the Taking of Anti-aromatases (AI) in Patients With Non-metastatic Breast Cancer
Brief Title: Evaluation of the Efficacy of a Homeopathic Protocol in Patients With Non-metastatic Breast Cancer
Acronym: ARHOMA2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Jean-Godinot (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-A01019-46
Record Dates: First submitted 2019-04-04; First posted 2020-05-29 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Breast Cancer Female; Joint Pain
MeSH Terms: conditions — Arthralgia | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Groupe A with homéopathic treatment (Active Comparator): Conventional treatment : paracetamol (drug analgesic class1) + Homeopathic drug : Rhus toxicodendron 9 CH et Ruta graveolens 5 CH
  Interventions: Drug: Rhus toxicodendron 9 CH + Ruta graveolens 5 CH (Homeopathic Granules); Other: paracetamol (drug analgesic class1)
- Groupe B without homeopathic treatment (Sham Comparator): Conventional treatment : paracetamol (drug analgesic class1)
  Interventions: Other: paracetamol (drug analgesic class1)

INTERVENTIONS:
Drug: Rhus toxicodendron 9 CH + Ruta graveolens 5 CH (Homeopathic Granules) — Rhus toxicodendron 9 CH + Ruta graveolens 5 CH
  Arms: Groupe A with homéopathic treatment
Other: paracetamol (drug analgesic class1) — paracetamol (drug analgesic class1)

SUMMARY:
Interventional, randomised, prospective, monocentric study

DETAILED DESCRIPTION:
Interventional, randomised, prospective, monocentric study

Primary objective :

Demonstrate the interest of the homeopathic Protocol to reduce the onset or aggravation of joint pain as a result of the taking of AI compared to conventional care

Secondary objective :

Compare between the two treatment groups:

* Evolution of joint pain
* Evolution of joint stiffness-rate of onset of pain and joint stiffness-delay in onset or aggravation of pain-evolution of the number of painful locations-evolution of the impact of pain on the quality of the sleep-consumption of permitted concomitant treatments (analgesics)
* Evolution of symptoms of hormonal deprivation-adherence to AI treatment
* Tolerance to AI
* Change seen by patients
* Stop rate and switch of AI-rate of recurrence of breast cancer

Describe in patients receiving homeopathic treatment:

* Adherence to homeopathic treatment
* Tolerance to homeopathic treatment
* Group A: Group of patients receiving conventional treatment (drug analgesic class 1) for joint pain + homeopathic treatment
* Group B: Group of patients receiving conventional treatment (drug analgesic class 1) for joint pain

Schedule :

* Inclusions start at: 01/09/2018
* End date of inclusions: 01/09/2021
* End date of follow-up: 23/03/2022
* Study report: 23/03/2023

ELIGIBILITY:
Inclusion Criteria:

* menopausal patient
* achieved histologically confirmed non-metastatic breast cancer with positive hormonal receptors
* starting an adjuvant anti-hormonal treatment with an AI
* patient benefiting from a social protection scheme
* patient mastering the French language -signature of free and informed consent -

Exclusion Criteria:

* patient whose treatment with chemotherapy or radiotherapy is ongoing or anticipated during the theoretical period of the study or patient who has completed her chemotherapy treatment within a period of less than 4 weeks prior to the inclusion visit
* patient with proven inflammatory rheumatism already diagnosed with rheumatoid arthritis, lupus, psoriatic rheumatism, ankylosing spondylitis -concomitant treatment with other complementary medicines (excepted Vitamin D), unless the treatment has been stable for at least 1 month.
* current treatment with narcotic drugs or corticosteroids
* patient with overexpressing breast cancer HER2

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2018-09-13 (Actual); Primary Completion 2021-08-27 (Actual); Study Completion 2022-03-23 (Actual)

PRIMARY OUTCOMES:
Evolution of the score of "most intense pain" during the first 3 months of treatment with AI | 3 months
  Evaluation comparing between the 2 groups the area under the most intense pain curve, measured each week during the first 3 months of AI treatment using the Brief Pain Inventory-Short Form (BPI-SF) scale (1 no disconfort up to 10 complet disconfort)

SECONDARY OUTCOMES:
Evolution of joint pain | 6 months
  variation of different pain scores on the Brief Pain Inventory-Short Form (BPI-SF) scale (1 no disconfort up to 10 complet disconfort) : pain severity score corresponding to the average of the 4 questions on pain intensity, and interference score corresponding to the average of the 7 questions on the impact of pain
Rate of onset of joint pain and stiffness | 3 months
  For pain, among patients who answered "no" to the first question of Brief Pain Inventory-Short Form (1 no disconfort up to 10 complet disconfort) to visit 1, percentage of patients who answered "Yes" to 3 months (visit 2)
Rate of onset of pain and joint stiffness | 3 months
  Percentage of patients for whom pain and / or stiffness have occurred.
Time of onset or aggravation of pain | 6 months
  time from which the "most severe pain" score has increased for at least 2 consecutive weeks since the Visit 1 score

CONTACTS AND LOCATIONS:
Overall Officials: PHILIPPE GUILBERT, Principal Investigator — Institut Jean-Godinot
Locations (1):
- Philippe GUILBERT, Reims, France

IPD SHARING:
Plan to Share IPD: No